CLINICAL TRIAL: NCT02290782
Title: TARGIT-C(Consolidation) Prospective Phase IV Study of Intraoperative Radiotherapy (IORT) in Patients With Small Breast Cancer
Brief Title: TARGIT-C(Consolidation) Prospective Phase IV Study of IORT in Patients With Small Breast Cancer
Acronym: TARGIT-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Elena Sperk, MD, Head, Clinical Trials Unit, Department of Radiation Oncology Mannheim, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARGIT C
Record Dates: First submitted 2014-10-30; First posted 2014-11-14 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: toxicity; outcome; TARGIT; quality of life; intraoperative radiotherapy (IORT)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm study: IORT +/- EBRT (risk adapted approach).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative radiotherapy (IORT) (Experimental): IORT (20Gy) as intervention will be given during breast conserving surgery. If risk factors (Tumor > 3.5 cm, lobular cancer, resection margin < 2 mm*, L1, pN+ mulitfocal/multicentric, EIC, negative hormone receptors) are present, external beam radiotherapy will be added.
  * In case of positive margins (<2 mm resection margin) a re-resection should be done
  Interventions: Radiation: Intraoperative radiotherapy (IORT)

INTERVENTIONS:
Radiation: Intraoperative radiotherapy (IORT) — The surgeon and radiation oncologist should choose the largest possible suitable applicator in order to ensure that the highest possible dose is delivered to the tumor bed tissue. A dose of 20 Gy at the surface of the applicator (in water) is prescribed by the radiation oncologist and delivered to the breast tissue. This takes approximately 20-50 minutes, depending on the size of the applicator.
  To minimize radiation dependent side effects the skin-applicator surface distance should be more than 5 mm.

SUMMARY:
This prospective, multicentric single arm phase IV study is based on the protocol of the international TARGIT-A and TARGIT-E study.

Patients ≥ 50 years with small, low-risk breast cancer who are operated but not irradiated show local relapse rates around 6% after 5 years. With adjuvant whole breast radiotherapy (WBRT) the local relapse rate drops to under 1% after 5 years under Tamoxifen (4).

It has been demonstrated (6, 9, 10) that the efficacy of radiation of the tumor bed only in a selected group can be non-inferior to WBRT.

The TARGIT C study should confirm the efficacy of a single dose of intraoperative radiotherapy (IORT) in a well selected group of patients with small breast cancer and absence of risk factors. In presence of risk factors postoperative WBRT will be added to complete the radiotherapeutic treatment according to international guidelines.

Endpoints are the local relapse rate (within 2 cm of the tumor bed), ipsilateral relapse, cancer-specific and overall survival and contralateral breast cancer as well as documentation of quality of life and cosmetic outcome.

The expected local relapse rates are 0.825/1.375% after 3/5 years, respectively. Discontinuation of the trial is scheduled if rates of local relapse rates rise to 1.55/2.4/4% after 1/3/5 years. Power calculations result in 387 patients with a calculated dropout and loss to follow-up rate of 10%, an alpha of 0.05 and a beta of 0.10. There will be only a pre-pathology stratum.

It is a pragmatic trial in which each participating centre has the option to modify entry criteria and criteria for WBRT according to this core protocol after consultation with the steering committee and local ethics committee (e.g. size, free margins). Only centers with access to the Intrabeam® system (Carl Zeiss) can recruit patients into the trial.

DETAILED DESCRIPTION:
1. Introduction

   Randomized studies provide evidence that concerning the overall survival breast conserving surgery (BCS) combined with postoperative radiotherapy is equally effective as modified mastectomy (1, 2, 3). Postoperative radiation decreases the local relapse rate (1, 2) highly significantly in comparison to BCS alone (3). The recent metaanalysis of the Early Breast Cancer Trialists Collaborative Group (EBCTCG (3)) show that the avoidance of 4 local relapses after 5 years can prevent one death in 15 years (4 to 1 rule).

   Several studies in the past demonstrated that complete omission of radiotherapy failed in terms of local tumor control. Fyles et al. (4) showed local relapse rates of 8% within a low risk group of patients with tumors of pathological stage T1/T2 and >50 years of age treated with BCS and antihormonal treatment (AHT). By adding postoperative whole breast radiation (WBRT) the rate of local relapse was reduced to 1% after 5 years. This effect was also seen in elderly patients with small tumors. Hughes et al. (5) observed low local relapse rates of 4% for patients treated with AHT only after BCS vs. 1% for patients with additional WBRT after 4 years, evaluating a low-risk group of patients with tumors < 2 cm and > 70 years of age. Apparently, all patients benefit from postoperative WBRT. However, due to the fact that 90% of all local relapses after breast conserving therapy are localized very close to the primary tumor, it might be possible to treat a selected group of patients with a relatively low risk of local recurrence with tumor bed irradiation only. Polgar et al. (6) provided evidence of the non-inferiority of accelerated partial breast irradiation (APBI) in comparison to WBRT in a small randomized trial. Very recently the TARGIT-A data (9, 10) reported a non-inferior efficacy of tumor bed irradiation with single dose intraoperative radiation (Intrabeam System, Carl Zeiss Oberkochen) compared to WBRT regarding local relapse.

   By using the Intrabeam System, the intraoperative radiotherapy (IORT) can be given during surgery with protection of the surrounding tissue while applying a biologically highly effective dose to the tissue adjacent to the tumor.

   Advantages of IORT are its high precision regarding beam application, its possibility of protection of the skin and the prevention of tumor cell proliferation during the time interval between breast conserving surgery and adjuvant WBRT as well as during fractionated WBRT.

   By manually positioning of the applicator in the tumor bed geographic miss is excluded and radiation of risk structures like the heart and lung can be avoided. Therefore, it is possible to give a high single fraction to the target and minimize relevant side effects.
2. Aim

The objective of this single armed phase IV study is to further investigate the efficacy of a single intraoperative radiotherapy treatment within low risk patients (≥ 50 years, cT1 and small cT2 (< 3.5 cm), cN0, cM0, invasive-ductal, hormone receptor positive) which is followed by WBRT only when risk factors are present.

The primary endpoint is the rate of local relapse (within 2 cm of the initial tumor); secondary endpoints are ipsi- or contralateral breast cancer, cancer specific and overall survival. Of further interest is the cosmetic outcome and Quality of Life.

Therefore, patients ≥ 50 years with small, histologically verified and hormone receptor positive invasive-ductal breast cancer (clinically cT1 or small T2 ≤ 3.5 cm) without risk factors (multifocality/- centricity, extensive intraductal component (EIC), lymph vessel invasion (L1), clinically positive lymph nodes) who receive BCS will be recruited.

After tumor resection with free margins > 1 mm the applicator will be exactly positioned in the tumor bed with a minimum distance to skin of 5 mm. The prescription dose will be 20 Gy to the surface of the applicator. The treatment times depend on the diameter of the applicator and can last up to 20-50 minutes. After radiation the applicator will be removed and the operation finished as usual. The biologic effectiveness of 20 Gy prescribed during the operation is equivalent to 70 Gy normo-fractionated irradiation according to radiobiological modelling.

If the final histopathological report provides evidence of a different histology or risk factors, such as an extensive intraductal component (EIC), lymph vessel invasion (L1), multifocality/-centricity or resection margins <2 mm, patients will receive a postoperative WBRT with 46 Gy (after a delay of at least 5 weeks). Depending on the lymph node status postoperative WBRT will be performed with 50 Gy (pN1) or WBRT including lymphatic drainage with 50 Gy (≥ pN2). A re-resection has to be performed in presence of insufficient free margins (e.g. tumor on ink, or margin < 2mm depending on local policy) and will be followed by WBRT with 50 Gy omitting the boost.

Cosmetic outcome and toxicity evaluation will be performed by chart (CTC and LENT-SOMA score) and standardized photo documentation.

For Quality of Life assessment the patients will complete two standardized and validated questionnaires developed by the EORTC (European Organisation for Research and Treatment of Cancer). The questionnaires include 53 questions and take approximately 10 minutes and will be filled out at clinic visits.

Therefore, a patient group including patients ≥ 50 years with a low-risk tumor profile will be treated in this single-arm study by intraoperative radiotherapy of the tumor bed only, using a well established method (Intrabeam System, Carl Zeiss Surgical, Oberkochen, Germany) in order to optimize radiotherapy treatment after breast conserving surgery in terms of local relapse, toxicity, overall survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified invasive-ductal breast cancer
* hormone receptor positive (if known)
* cT1 or small cT2 (≤ 3.5 cm) cN0 cM0
* ≥ 50 years of age
* informed consent
* compliance

Exclusion Criteria:

* extensive intraductal component (EIC)
* negative hormone receptor status
* multifocality /-centricity (mammography, breast ultrasound)
* lymph vessel invasion (L1)
* clinical signs of distant metastases or clinically suspicious lymph nodes
* other histology
* < 50 years
* missing informed consent or non-compliance
* bilateral breast cancer at the time of diagnosis
* known BCRA1/2 gene mutations (genetic testing not required)
* any exclusion criterion in the local centre´s treatment policy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer in females
Enrollment: 387 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local relapse | 5 years
  Local relapse rate within 2 cm of the tumor bed

SECONDARY OUTCOMES:
Ipsi- or contralateral breast cancer | 5 years
  Ipsi- or contralateral breast cancer
Survival | 5 years
  Breast cancer related and overall survival
Toxicity (CTC, LENT SOMA) | 5 years
  Cosmetic outcome, acute and late toxicity measured by CTC Score V5 and LENT SOMA scale (fibrosis, telangiectasia, edema arm, edema breast, ulceration, hyperpigmentation, pain, retraction
General QoL and breast specific QoL (EORTC QLQ C30 + BR23) | 5 years
  measured by EORTC QLQ C30 and BR23 questionnaires; longitudinal analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sperk, MD, Principal Investigator — department of radiation oncology
Locations (4):
- France (2):
  - Institut régional du Cancer de Montpellier, Montpellier
  - IUCT, Toulouse, Toulouse
- Germany (2):
  - Klinikum Kassel, Kassel
  - Department of Radiotherapy University Hospital Mannheim, Mannheim

REFERENCES:
- [Background] Fisher B, Anderson S, Redmond CK, Wolmark N, Wickerham DL, Cronin WM. Reanalysis and results after 12 years of follow-up in a randomized clinical trial comparing total mastectomy with lumpectomy with or without irradiation in the treatment of breast cancer. N Engl J Med. 1995 Nov 30;333(22):1456-61. doi: 10.1056/NEJM199511303332203. PMID 7477145
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Fyles AW, McCready DR, Manchul LA, Trudeau ME, Merante P, Pintilie M, Weir LM, Olivotto IA. Tamoxifen with or without breast irradiation in women 50 years of age or older with early breast cancer. N Engl J Med. 2004 Sep 2;351(10):963-70. doi: 10.1056/NEJMoa040595. PMID 15342804
- [Background] Hughes KS, Schnaper LA, Berry D, Cirrincione C, McCormick B, Shank B, Wheeler J, Champion LA, Smith TJ, Smith BL, Shapiro C, Muss HB, Winer E, Hudis C, Wood W, Sugarbaker D, Henderson IC, Norton L; Cancer and Leukemia Group B; Radiation Therapy Oncology Group; Eastern Cooperative Oncology Group. Lumpectomy plus tamoxifen with or without irradiation in women 70 years of age or older with early breast cancer. N Engl J Med. 2004 Sep 2;351(10):971-7. doi: 10.1056/NEJMoa040587. PMID 15342805
- [Background] Polgar C, Fodor J, Major T, Nemeth G, Lovey K, Orosz Z, Sulyok Z, Takacsi-Nagy Z, Kasler M. Breast-conserving treatment with partial or whole breast irradiation for low-risk invasive breast carcinoma--5-year results of a randomized trial. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):694-702. doi: 10.1016/j.ijrobp.2007.04.022. Epub 2007 May 25. PMID 17531400
- [Background] Kraus-Tiefenbacher U, Bauer L, Kehrer T, Hermann B, Melchert F, Wenz F. Intraoperative radiotherapy (IORT) as a boost in patients with early-stage breast cancer -- acute toxicity. Onkologie. 2006 Mar;29(3):77-82. doi: 10.1159/000091160. Epub 2006 Mar 3. PMID 16514267
- [Background] Kraus-Tiefenbacher U, Bauer L, Scheda A, Fleckenstein K, Keller A, Herskind C, Steil V, Melchert F, Wenz F. Long-term toxicity of an intraoperative radiotherapy boost using low energy X-rays during breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2006 Oct 1;66(2):377-81. doi: 10.1016/j.ijrobp.2006.05.042. Epub 2006 Aug 2. PMID 16887294
- [Background] Vaidya JS, Joseph DJ, Tobias JS, Bulsara M, Wenz F, Saunders C, Alvarado M, Flyger HL, Massarut S, Eiermann W, Keshtgar M, Dewar J, Kraus-Tiefenbacher U, Sutterlin M, Esserman L, Holtveg HM, Roncadin M, Pigorsch S, Metaxas M, Falzon M, Matthews A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy versus whole breast radiotherapy for breast cancer (TARGIT-A trial): an international, prospective, randomised, non-inferiority phase 3 trial. Lancet. 2010 Jul 10;376(9735):91-102. doi: 10.1016/S0140-6736(10)60837-9. PMID 20570343
- [Background] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Background] Vaidya JS, Bulsara M, Baum M, Wenz F, Massarut S, Pigorsch S, Alvarado M, Douek M, Saunders C, Flyger HL, Eiermann W, Brew-Graves C, Williams NR, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Corica T, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Le Blanc-Onfroy M, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McCready D, Hoefer R, Kelemen P, Petralia G, Falzon M, Joseph DJ, Tobias JS. Long term survival and local control outcomes from single dose targeted intraoperative radiotherapy during lumpectomy (TARGIT-IORT) for early breast cancer: TARGIT-A randomised clinical trial. BMJ. 2020 Aug 19;370:m2836. doi: 10.1136/bmj.m2836. PMID 32816842